CLINICAL TRIAL: NCT02745821
Title: Coronary Physiology and Its Relationship to Anatomy in Patients With Diabetes Mellitus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20150876
Record Dates: First submitted 2016-04-04; First posted 2016-04-20 (Estimated); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus; Coronary Artery Disease
Keywords: coronary flow reserve; fractional flow reserve; diabetes mellitus; coronary artery disease; percutaneous coronary intervention; coronary physiology; index of microcirculatory resistance
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Coronary physiology (Experimental): Non-target and target vessels of patients with diabetes mellitus referred for PCI will be assessed for FFR, CFR and IMR. Intravenous adenosine at 140 micrograms/kg/min will be used to induce maximal hyperemia.
  Interventions: Device: Pressure Wire Certus, St. Jude Medical, USA

INTERVENTIONS:
Device: Pressure Wire Certus, St. Jude Medical, USA — FFR. CFR and IMR will be measured using the Pressure Wire Certus, St. Jude Medical, USA in target and non-target vessels. Changes in FFR, CFR and IMR post PCI of target vessels will also be recorded.

SUMMARY:
Comprehensive assessment of coronary physiology (fractional flow reserve (FFR), coronary flow reserve (CFR) and index of microcirculatory resistance (IMR)) in patients with diabetes mellitus and coronary artery disease (CAD).

DETAILED DESCRIPTION:
Background:

There is currently no data on invasive measurement of FFR, CFR and IMR in patients with diabetes mellitus. Studies such as RIPCORD has shown that using coronary angiography alone to guide revascularization strategy may be flawed in a significant proportion of patients.

Patients with diabetes mellitus are more likely to have diffuse CAD and microvascular disease. Current recommendation of invasive physiological assessment to guide percutaneous coronary intervention (PCI) is limited to FFR alone. This can be misleading in diffuse coronary artery disease and microvascular disease as both conditions are associated with higher FFR. The proportion of vessels which show discordance between FFR and CFR consistent with diffuse CAD and/or microvascular disease in patients has been shown to be as high as 30% in a study not exclusive to diabetics.

This is a pilot study of 50 patients referred for PCI based on angiographic stenosis of ≥50%. Comprehensive physiological assessment will be undertaken in target and non-target vessels to determine the prevalence of discordant FFR and CFR consistent with diffuse CAD and/or microvascular dysfunction in diabetics.

Methods:

1. Patients will receive an information sheet after initial invitation to participate in the study.
2. Written informed consent will be obtained.
3. Patients will undergo invasive assessment of FFR, CFR and IMR in non-target vessels.
4. An optical coherence tomography (OCT) study will be performed to correlate physiological parameters with intravascular imaging for diffuse atheromatous disease.
5. Patients will then undergo OCT and invasive assessment of FFR, CFR and IMR in the target vessel pre and post PCI.
6. Any change in FFR, CFR and IMR post PCI will be recorded.
7. All physiological parameters will be measured using the pressure wire from St. Jude Medical, USA (currently, Certus). Results will be grouped according to 4 possible permutations of FFR and CFR.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with angina and/or evidence of myocardial ischemia (includes ACS patients but not STEMI)
* Willing and able to provide informed, written consent
* Diabetic patients with clinically indicated, abnormal PET scan
* Single or double vessel disease with coronary stenosis ≥50% referred for PCI

Exclusion Criteria:

* Significant left main stenosis ≥50% and/or triple vessel disease referred for CABG
* Recent STEMI (<5 days)
* Previous CABG
* LVEF ≤ 30% or cardiogenic shock
* Complex coronary anatomy preventing FFR/CFR measurement

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06; Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of number of vessels fulfilling each of 4 permutations of fractional flow reserve (FFR) and coronary flow reserve (CFR) ie FFR ≤0.80 CFR ≥2.0, FFR ≤0.80 CFR <2.0, FFR >0.80 CFR ≥2.0 and FFR >0.80 CFR <2.0. | Duration of procedure in the catheterization laboratory ie 1 day
  This is primarily an observational pilot study where coronary physiology is obtained at the time of the percutaneous coronary intervention (PCI) of the target vessel.

SECONDARY OUTCOMES:
Change in FFR in target vessel | Baseline and post PCI
  FFR will be measured pre and post PCI of target vessel
Change in CFR in target vessel | Baseline and post PCI
  CFR will be measured pre and post PCI of target vessel
Change in index of microvascular resistance (IMR) in target vessel | Baseline and post PCI
  IMR will be measured pre and post PCI of target vessel

CONTACTS AND LOCATIONS:
Overall Officials: Aun-Yeong Chong, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Curzen N, Rana O, Nicholas Z, Golledge P, Zaman A, Oldroyd K, Hanratty C, Banning A, Wheatcroft S, Hobson A, Chitkara K, Hildick-Smith D, McKenzie D, Calver A, Dimitrov BD, Corbett S. Does routine pressure wire assessment influence management strategy at coronary angiography for diagnosis of chest pain?: the RIPCORD study. Circ Cardiovasc Interv. 2014 Apr;7(2):248-55. doi: 10.1161/CIRCINTERVENTIONS.113.000978. Epub 2014 Mar 18. PMID 24642999
- [Background] Echavarria-Pinto M, Escaned J, Macias E, Medina M, Gonzalo N, Petraco R, Sen S, Jimenez-Quevedo P, Hernandez R, Mila R, Ibanez B, Nunez-Gil IJ, Fernandez C, Alfonso F, Banuelos C, Garcia E, Davies J, Fernandez-Ortiz A, Macaya C. Disturbed coronary hemodynamics in vessels with intermediate stenoses evaluated with fractional flow reserve: a combined analysis of epicardial and microcirculatory involvement in ischemic heart disease. Circulation. 2013 Dec 17;128(24):2557-66. doi: 10.1161/CIRCULATIONAHA.112.001345. Epub 2013 Oct 18. PMID 24141255